CLINICAL TRIAL: NCT01192022
Title: A Randomized, Open Label, Parallel-group, Multi-center Trial to Compare the Efficacy and Safety of TachoSil® Versus Surgicel® Original for the Secondary Treatment of Local Bleeding in Adult and Pediatric Patients Undergoing Hepatic Resection Surgery
Brief Title: TachoSil® Versus Surgicel® Original for the Secondary Treatment of Local Bleeding in Adult and Pediatric Patients Undergoing Hepatic Resection Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TC-2402-040-SP; U1111-1130-9121 (Registry Identifier: WHO)
Record Dates: First submitted 2010-08-27; First posted 2010-08-31 (Estimated); Results first posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-10

CONDITIONS: Hemorrhage
Keywords: Liver resection; Liver transplantation; Liver surgery; Secondary hemostasis
MeSH Terms: conditions — Hemorrhage | interventions — TachoSil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TachoSil® (Active Comparator): TachoSil® absorbable patches, applied topically, once, intraoperatively to stop bleeding. The number of patches used was determined by the surgeon based on the size of the wound. If bleeding did not stop after 5 minutes treatment was repeated.
  Interventions: Biological: TachoSil®
- Surgicel® Original (Active Comparator): Surgicel® Original absorbable patches, applied topically, once, intraoperatively to stop bleeding. The number of patches used was determined by the surgeon based on the size of the wound. If bleeding did not stop after 5 minutes treatment was repeated.
  Interventions: Device: Surgicel® Original

INTERVENTIONS:
Biological: TachoSil® — Intraoperative application as secondary hemostatic treatment
  Arms: TachoSil®
Device: Surgicel® Original — Intraoperative application as secondary hemostatic treatment
  Arms: Surgicel® Original

SUMMARY:
The efficacy and safety of TachoSil® as secondary hemostatic treatment in hepatic resection surgery will be compared to the standard USA licensed hemostatic agent, Surgicel® Original. Hemostatic efficacy will be evaluated intraoperatively after application of randomized treatment.

ELIGIBILITY:
Inclusion Criteria:

* Resection of at least the equivalent tissue volume of 1 anatomical segment of the liver
* Minor to moderate (oozing/diffuse) bleeding from the resection area persisting after conventional resection procedure and primary control of arterial pulsating bleeding or major venous hemorrhage by sutures, ligations, clips, vascular stapler, point electrocautery or focal radiofrequency ablation
* Need for additional supportive hemostatic treatment
* Expected ability to lightly press the trial treatment to the liver resection wound for 3 minutes

Exclusion Criteria:

* Indication for emergency surgery
* Known coagulopathy (as judged relevant by the investigator)
* Known or suspected hypersensitivity to any ingredient of the investigational medicinal products (e.g. human fibrinogen, human thrombin and/or collagen of any origin)
* Patient unwilling to receive blood products
* Known current alcohol or drug abuse
* Pregnancy, breastfeeding, no use of acceptable contraceptive method in females of childbearing potential
* Dry surgical field of the targeted application area
* Occurrence of any serious surgical complication
* Disseminated intravascular coagulopathy (DIC), i.e. microvascular bleeding
* Application of topical hemostatic material on the liver resection wound
* Radiofrequency precoagulation of the liver resection wound except focal radiofrequency ablation of vessels as primary hemostatic treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2010-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (17):
- United States (17):
  - Los Angeles, California
  - Washington D.C., District of Columbia
  - Chicago, Illinois
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Burlington, Massachusetts
  - St Louis, Missouri
  - Newark, New Jersey
  - New York, New York
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Charlottesville, Virginia
  - Madison, Wisconsin

REFERENCES:
- [Derived] Genyk Y, Kato T, Pomposelli JJ, Wright JK Jr, Sher LS, Tetens V, Chapman WC. Fibrin Sealant Patch (TachoSil) vs Oxidized Regenerated Cellulose Patch (Surgicel Original) for the Secondary Treatment of Local Bleeding in Patients Undergoing Hepatic Resection: A Randomized Controlled Trial. J Am Coll Surg. 2016 Mar;222(3):261-8. doi: 10.1016/j.jamcollsurg.2015.12.007. Epub 2015 Dec 18. PMID 26776356

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants took part in the study at 19 investigative sites in the United States from 31 August 2010 to 07 November 2012. Pediatric participants took part in the study at 5 investigative sites in the United States from 09 March 2012 to 03 May 2013.
Pre-assignment Details: Adult and pediatric participants were enrolled equally in 1 of 2 treatment groups, TachoSil or Surgicel Original, applied once or twice if needed intraoperatively during a 10-minute observation period, or until hemostasis was obtained. Pediatric enrollment continued in an extension phase where all participants were allocated to TachoSil.
Groups:
- TachoSil® (Adult Participants); TachoSil® (Pediatric Participants); TachoSil® Extension Analysis Set (Pediatric Participants): TachoSil® absorbable patches, applied topically, once, intraoperatively to stop bleeding. The number of patches used was determined by the surgeon based on the size of the wound. If bleeding did not stop after 5 minutes treatment was repeated.
- Surgicel® Original (Adult Participants); Surgicel® Original (Pediatric Participants): Surgicel® Original absorbable patches, applied topically, once, intraoperatively to stop bleeding. The number of patches used was determined by the surgeon based on the size of the wound. If bleeding did not stop after 5 minutes treatment was repeated.
Period: Overall Study
Arm/Group | TachoSil® (Adult Participants) | Surgicel® Original (Adult Participants) | TachoSil® (Pediatric Participants) | Surgicel® Original (Pediatric Participants) | TachoSil® Extension Analysis Set (Pediatric Participants)
Started | 114 | 110 | 8 | 9 | 12
Safety Population-Received Treatment | 114 | 109 | 8 | 9 | 12
Completed | 101 | 99 | 7 | 7 | 11
Not Completed | 13 | 11 | 1 | 2 | 1
Not completed — Withdrawal of Consent | 3 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 2 | 1 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Fatal Adverse Event | 4 | 6 | 0 | 0 | 1
Not completed — Physician withdrew-patient hardship | 1 | 0 | 0 | 0 | 0
Not completed — Patient too sick from chemotherapy | 0 | 1 | 0 | 0 | 0
Not completed — Patient needed surgery | 0 | 1 | 0 | 0 | 0
Not completed — Parents did not allow all follow up | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The TachoSil pediatric arm includes pediatric participants who were randomized to receive TachoSil, in addition to pediatric participants who were allocated to receive TachoSil via the extension phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | TachoSil® (Adult Participants) | Surgicel® Original (Adult Participants) | TachoSil® (Pediatric Participants) | Surgicel® Original (Pediatric Participants) | Total
Number analyzed (Participants) | 114 | 110 | 20 | 9 | 253
Age, Continuous [Mean (Standard Deviation); unit: years] — Adult Participants
  years | 58.4 (13.69) | 57.8 (14.27) | NA (NA) — Pediatric population reported separately. | NA (NA) — Pediatric population reported separately | 58.1 (13.95)
Age, Continuous [Mean (Standard Deviation); unit: years] — Pediatric Participants
  years | NA (NA) — Adult participants reported separately. | NA (NA) — Adult participants reported separately. | 4.58 (4.716) | 3.77 (5.107) | 4.33 (4.764)
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.4 (13.69) | 57.8 (14.27) | 4.58 (4.716) | 3.77 (5.107) | NA (NA) — Total Mean and SD not calculated for the 4 Arms combined.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 51 | 10 | 5 | 120
  Male | 60 | 59 | 10 | 4 | 133
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 93 | 87 | 16 | 7 | 203
  Asian | 6 | 10 | 2 | 1 | 19
  Black or African American | 9 | 10 | 1 | 0 | 20
  Mixed race | 2 | 0 | 0 | 0 | 2
  Other | 4 | 3 | 1 | 1 | 9
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 8 | 7 | 4 | 2 | 21
  Non-Hispanic/Non-Latino | 98 | 98 | 14 | 6 | 216
  Unknown | 8 | 5 | 2 | 1 | 16
Age, Categorical: Adult Population [Number; unit: participants]
  ≤65 years | 81 | 76 | NA — Pediatric age is reported separately. | NA — Pediatric age is reported separately. | NA — Total not calculated because data are not available (NA) in one or more arms.
  >65 years | 33 | 34 | NA — Pediatric age is reported separately. | NA — Pediatric age is reported separately. | NA — Total not calculated because data are not available (NA) in one or more arms.
Age, Categorical: Pediatric Population [Number; unit: participants]
  0-23 months | NA — Adult age is reported separately. | NA — Adult age is reported separately. | 9 | 5 | NA — Total not calculated because data are not available (NA) in one or more arms.
  2-11 years | NA — Adult age is reported separately. | NA — Adult age is reported separately. | 8 | 3 | NA — Total not calculated because data are not available (NA) in one or more arms.
  12-16 years | NA — Adult age is reported separately. | NA — Adult age is reported separately. | 3 | 1 | NA — Total not calculated because data are not available (NA) in one or more arms.
Height: Adult Population [Mean (Standard Deviation); unit: cm] | 169.30 (9.927) | 170.33 (9.929) | NA (NA) — Pediatric height is reported separately. | NA (NA) — Pediatric height is reported separately. | 169.81 (9.919)
Height: Pediatric Population [Mean (Standard Deviation); unit: cm] — Number of participants for whom pediatric height data were available were 19 and 7 in each treatment arm, respectively.
  cm | NA (NA) — Adult height is reported separately. | NA (NA) — Adult height is reported separately. | 96.36 (36.588) | 77.39 (24.650) | 91.25 (34.400)
Weight: Adult Population [Mean (Standard Deviation); unit: kg] | 80.46 (16.968) | 79.03 (18.545) | NA (NA) — Pediatric weight is reported separately. | NA (NA) — Pediatric weight is reported separately. | 79.75 (17.737)
Weight: Pediatric Population [Mean (Standard Deviation); unit: kg] — Number of participants for whom pediatric weight data were available were 19 and 8 in each treatment arm, respectively.
  kg | NA (NA) — Adult weight is reported separately. | NA (NA) — Adult weight is reported separately. | 19.48 (17.783) | 11.11 (7.963) | 17.00 (15.848)
Body Mass Index (BMI): Adult Population [Mean (Standard Deviation); unit: kg/m^2] | 28.09 (5.521) | 27.16 (5.653) | NA (NA) — Pediatric BMI is reported separately. | NA (NA) — Pediatric BMI is reported separately. | 27.64 (5.593)
Body Mass Index (BMI): Pediatric Population [Mean (Standard Deviation); unit: kg/m^2] — Number of participants for whom pediatric BMI data were available were 19 and 7 in each treatment arm, respectively.
  kg/m^2 | NA (NA) — Adult BMI is reported separately. | NA (NA) — Adult BMI is reported separately. | 17.49 (3.103) | 16.57 (2.637) | 17.24 (2.962)
Fertility Status: Adult Population [Number; unit: participants]
  Menstrual | 6 | 5 | NA — Fertility status data was not collected for the pediatric population. | NA — Fertility status data was not collected for the pediatric population. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Postmenstrual | 26 | 24 | NA — Fertility status data was not collected for the pediatric population. | NA — Fertility status data was not collected for the pediatric population. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Surgically sterile | 22 | 22 | NA — Fertility status data was not collected for the pediatric population. | NA — Fertility status data was not collected for the pediatric population. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Not applicable | 60 | 59 | NA — Fertility status data was not collected for the pediatric population. | NA — Fertility status data was not collected for the pediatric population. | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Intraoperative Hemostasis at Target Bleeding Site Within 3 Minutes
Description: 3 Minutes after the patch was applied to the target bleeding area, the area was observed to see if the bleeding stopped.
Time Frame: within 3 minutes
Population: Full Analysis set included all randomized participants analyzed according to the treatment assigned.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TachoSil® (Adult Participants) | Surgicel® Original (Adult Participants) | TachoSil® (Pediatric Participants) | Surgicel® Original (Pediatric Participants) | TachoSil® Extension Analysis Set (Pediatric Participants)
Number analyzed (Participants) | 114 | 110 | 8 | 9 | 12
percentage of participants | 80.7 [72.3 to 87.5] | 50.0 [40.3 to 59.7] | 87.5 [47.3 to 99.7] | 44.4 [13.7 to 78.8] | 83.3 [51.6 to 97.9]
Statistical Analysis 1: Comparison: TachoSil® (Adult Participants) vs Surgicel® Original (Adult Participants); Test type: Superiority or Other; p < 0.001, Regression, Logistic — Logistic regression model with treatment and pooled center as factors; Odds Ratio (OR) = 4.87, 95% CI 2-sided [2.55 to 9.29], Standard Error of Mean 1.60

2. Secondary Outcome: Percentage of Participants With Intraoperative Hemostasis at Target Bleeding Site Within 5 Minutes
Description: 3, 4 and 5 minutes after the patch was applied to the target bleeding area, the area was observed to see if the bleeding stopped.
Time Frame: within 5 minutes
Population: Full Analysis set included all randomized participants analyzed according to the treatment assigned.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TachoSil® (Adult Participants) | Surgicel® Original (Adult Participants) | TachoSil® (Pediatric Participants) | Surgicel® Original (Pediatric Participants) | TachoSil® Extension Analysis Set (Pediatric Participants)
Number analyzed (Participants) | 114 | 110 | 8 | 9 | 12
percentage of participants | 94.7 [88.9 to 98.0] | 76.4 [67.3 to 83.9] | 87.5 [47.3 to 99.7] | 77.8 [40.0 to 97.2] | 100.00 [73.5 to 100.0]

3. Secondary Outcome: Time to Intraoperative Hemostasis at Target Bleeding Site
Description: The target bleeding area was observed at 3, 4, 5, 8, 9, and 10 minutes after the patch was applied to see if the bleeding stopped, and time in minutes until bleeding stopped was recorded.
Time Frame: 10 minutes
Population: Full Analysis set included all randomized participants analyzed according to the treatment assigned.
Measure: Median (Full Range); unit: minutes
Arm/Group | TachoSil® (Adult Participants) | Surgicel® Original (Adult Participants) | TachoSil® (Pediatric Participants) | Surgicel® Original (Pediatric Participants) | TachoSil® Extension Analysis Set (Pediatric Participants)
Number analyzed (Participants) | 114 | 110 | 8 | 9 | 12
minutes | 3.0 [3.0 to 10.0] | 3.0 [3.0 to 28.0] | 3.0 [3.0 to 8.0] | 3.5 [3.0 to 8.0] | 3.0 [3.0 to 5.0]

ADVERSE EVENTS:
Description: The Safety Population included all enrolled participants who received treatment.
  At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TachoSil® (Adult Participants) | Surgicel® Original (Adult Participants) | TachoSil® (Pediatric Participants) | Surgicel® Original (Pediatric Participants)
Serious Adverse Events (participants affected / at risk) | 44/114 | 54/109 | 12/20 | 4/9
Other Adverse Events (participants affected / at risk) | 92/114 | 83/109 | 19/20 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TachoSil® (Adult Participants) (N=114) | Surgicel® Original (Adult Participants) (N=109) | TachoSil® (Pediatric Participants) (N=20) | Surgicel® Original (Pediatric Participants) (N=9)
Atrial fibrillation (Cardiac disorders) | 2 | 5 | 0 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 3 | 4 | 0 | 1
Abdominal abscess (Infections and infestations) | 3 | 2 | 0 | 0
Postoperative wound infection (Infections and infestations) | 3 | 0 | 0 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 4 | 7 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 3 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 2 | 2
Clostridium difficile colitis (Infections and infestations) | 1 | 2 | 2 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 2 | 1 | 0
Klebsiella infection (Infections and infestations) | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Bundle branch block right (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Syringomyelia (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Device occlusion (General disorders) | 0 | 1 | 0 | 0
Hernia obstructive (General disorders) | 0 | 1 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Biloma (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Hepatic ischaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Infectious peritonitis (Infections and infestations) | 2 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 2 | 1 | 0 | 0
Wound infection (Infections and infestations) | 2 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 2 | 0 | 0
Clostridial infection (Infections and infestations) | 1 | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Haematoma infection (Infections and infestations) | 1 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Subdiaphragmatic abscess (Infections and infestations) | 1 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Peritoneal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative abscess (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0
Wound abscess (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative adhesion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Antibiotic resistant Staphylococcus test positive (Investigations) | 0 | 1 | 0 | 0
False positive investigation result (Investigations) | 0 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hepatic neoplasm malignant recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colorectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 2 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 0 | 0
Urethral haemorrhage (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Activities of daily living impaired (Social circumstances) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 0 | 0
Shock (Vascular disorders) | 0 | 1 | 0 | 0
Disseminated intravasular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Catheter site swelling (General disorders) | 0 | 0 | 1 | 0
Hepatic artery thrombosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatic necrosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Alpha haemolytic streptococcal infection (Infections and infestations) | 0 | 0 | 1 | 0
Enterobacter infection (Infections and infestations) | 0 | 0 | 1 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 1 | 0
Mycobacterium abscessus infection (Infections and infestations) | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0
Stenotrophomonas infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Viraemia (Infections and infestations) | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 0 | 1
Anastomotic complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Incision site haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Exsanguination (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TachoSil® (Adult Participants) (N=114) | Surgicel® Original (Adult Participants) (N=109) | TachoSil® (Pediatric Participants) (N=20) | Surgicel® Original (Pediatric Participants) (N=9)
Anaemia (Blood and lymphatic system disorders) | 26 | 23 | 6 | 2
Neutropenia (Blood and lymphatic system disorders) | 5 | 3 | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 8 | 10 | 0 | 1
Tachycardia (Cardiac disorders) | 11 | 17 | 3 | 2
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 9 | 8 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 12 | 4 | 2 | 0
Constipation (Gastrointestinal disorders) | 28 | 31 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 13 | 19 | 2 | 0
Vomiting (Gastrointestinal disorders) | 15 | 15 | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 10 | 9 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 3 | 4 | 1 | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 3 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 3 | 1 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 4 | 10 | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 35 | 29 | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 2 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 13 | 10 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 6 | 4 | 0 | 0
Pyrexia (General disorders) | 16 | 22 | 8 | 3
Catheter site haematoma (General disorders) | 0 | 0 | 1 | 0
Fibrosis (General disorders) | 2 | 1 | 1 | 0
Oedema (General disorders) | 0 | 4 | 1 | 0
Oedema peripheral (General disorders) | 16 | 16 | 1 | 0
Generalised oedema (General disorders) | 1 | 1 | 0 | 1
Fatigue (General disorders) | 8 | 14 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 3 | 1 | 1 | 0
Hepatic vein stenosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Portal vein stenosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Venoocclusive liver disease (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 19 | 10 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Liver transplant rejection (Immune system disorders) | 0 | 0 | 1 | 0
Transplant rejection (Immune system disorders) | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1
Human herpesvirus 6 infection (Infections and infestations) | 0 | 0 | 2 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Clostridial infection (Infections and infestations) | 2 | 1 | 1 | 0
Epstein-Barr viraemia (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 1 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 1
Febrile infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 9 | 4 | 1 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 5 | 6 | 2 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hepatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Inadequate analgesia (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0
Procedural hypertension (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Transaminases increased (Investigations) | 4 | 2 | 2 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 1 | 0
Coagulation time prolonged (Investigations) | 1 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 1 | 0 | 1 | 0
Urine output decreased (Investigations) | 4 | 2 | 1 | 0
White blood cell count increased (Investigations) | 2 | 6 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 12 | 10 | 2 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1
Fluid imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 12 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 17 | 24 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 3 | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 18 | 8 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 4 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 14 | 9 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 7 | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 7 | 7 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 7 | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 5 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 5 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 5 | 5 | 0 | 1
Anxiety (Psychiatric disorders) | 4 | 3 | 1 | 0
Emotional distress (Psychiatric disorders) | 0 | 0 | 1 | 0
Emotional poverty (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 7 | 7 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 7 | 6 | 0 | 0
Dysuria (Renal and urinary disorders) | 2 | 1 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 5 | 4 | 1 | 0
Ketonuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Oliguria (Renal and urinary disorders) | 12 | 5 | 0 | 0
Urinary retention (Renal and urinary disorders) | 9 | 3 | 0 | 0
Scrotal swelling (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 17 | 18 | 2 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 22 | 13 | 1 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 13 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 8 | 0 | 1
Hypertension (Vascular disorders) | 14 | 10 | 3 | 1
Hypotension (Vascular disorders) | 22 | 20 | 3 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.